CLINICAL TRIAL: NCT00273780
Title: HAART Adherence Interventions in Africa: An RCT
Brief Title: Highly Active Antiretroviral Therapy (HAART) Adherence Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 29936-G; 1K23AI065222-01 (NIH); 5K23AI065222-02 (NIH)
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: HIV Infections
Keywords: Patient compliance
MeSH Terms: conditions — HIV Infections; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Adherence counseling (Active Comparator)
  Interventions: Behavioral: Adherence counseling
- Alarm device (Active Comparator)
  Interventions: Device: Alarm device
- Counseling and alarm (Active Comparator): Participants in this arm will receive both education counseling and a pocket alarm device.
  Interventions: Behavioral: Adherence counseling; Device: Alarm device
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Adherence counseling — Three adherence counseling sessions will be given to participants in the trial. Two sessions will occur prior to initiation of antiretroviral medications and one session will be given one month after drug administration.
  Arms: Adherence counseling; Counseling and alarm
Device: Alarm device — This pocket alarm device will be set to ring at designated times during the day that the participant should take their antiretroviral medication.
  Other Names: ALRT Med Reminder PC200
  Arms: Alarm device; Counseling and alarm

SUMMARY:
This study proposes a 4-armed factorial randomized clinical trial in Nairobi, Kenya to determine the effect of cognitive and behavioral interventions on HAART adherence.

DETAILED DESCRIPTION:
The study will be a prospective randomized clinical control trial among HIV-1 seropositive adult participants beginning HAART (highly active antiretroviral therapy) for the first time. Patients who are eligible to be initiated on HAART at the UW/Coptic Hope Center for Infectious Diseases will be referred for enrollment. Eligible patients who are referred will learn about the study and be invited to enroll after signing a written informed consent.

Study participants will be randomized to one of four arms:educational counseling, a pocket alarm device, both education and alarm, or neither. Participants will be followed in the study for 1 ½ years after enrollment and randomization. Participants will return to clinic every month to pick up a renewal of their antiretroviral prescriptions at which time pill counts will be performed. During follow-up visits, blood will be drawn and stored for CD4 counts and HIV-1 viral analyses.

Within this trial, the study also proposes to identify sociodemographic and spatial correlates of adherence. The study hypothesizes that educational counseling and medication alarm devices may significantly improve adherence, and that poor adherence may be associated with low socioeconomic standing, increased mobility, and distance from clinic.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must qualify for HAART treatment by World Health Organization (WHO) criteria (Clinical Stage IV disease) and/or CD4 count of less than 200 and plan to start HAART therapy.
* Must be above 18 years of age
* Must be HAART treatment-naïve
* Must agree to home visits, and plan to live in Kenya for at least two years.

Exclusion Criteria:

* Individuals who are mentally incompetent or are pregnant are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2006-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Pill count | 18 months

SECONDARY OUTCOMES:
CD4 count | 18 months
HIV-1 viral load | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Chung, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Hope Center for Infectious Diseases, Nairobi, Kenya

REFERENCES:
- [Derived] Marson KG, Tapia K, Kohler P, McGrath CJ, John-Stewart GC, Richardson BA, Njoroge JW, Kiarie JN, Sakr SR, Chung MH. Male, mobile, and moneyed: loss to follow-up vs. transfer of care in an urban African antiretroviral treatment clinic. PLoS One. 2013 Oct 24;8(10):e78900. doi: 10.1371/journal.pone.0078900. eCollection 2013. PMID 24205345
- [Derived] Chung MH, Richardson BA, Tapia K, Benki-Nugent S, Kiarie JN, Simoni JM, Overbaugh J, Attwa M, John-Stewart GC. A randomized controlled trial comparing the effects of counseling and alarm device on HAART adherence and virologic outcomes. PLoS Med. 2011 Mar;8(3):e1000422. doi: 10.1371/journal.pmed.1000422. Epub 2011 Mar 1. PMID 21390262